CLINICAL TRIAL: NCT00883935
Title: Phase I, Open Label, Randomized, Drug-Drug Interaction Study in Healthy Subjects to Investigate the Effects of Co-Administered Atazanavir/Ritonavir (300mg/100mg) or Atazanavir 400mg Administered Once Daily on the Steady-State Plasma Pharmacokinetics of GSK1349572 30mg Administered Once Daily
Brief Title: GSK1349572 Drug Interaction Study With Atazanavir/Ritonavir and Atazanavir
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Shionogi (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 111854
Record Dates: First submitted 2009-04-16; First posted 2009-04-20 (Estimated); Last update posted 2009-06-22 (Estimated); Status verified 2009-06

CONDITIONS: Healthy Volunteer
Keywords: GSK1349572; Atazanavir; Ritonavir; Reyataz; Norvir; healthy; pharmacokinetic
MeSH Terms: interventions — dolutegravir; Atazanavir Sulfate; Ritonavir

ARMS (2):
- Sequence 2 (Experimental): In the first treatment period, all subjects will receive GSK1349572 30mg q24h for 5 days (treatment A). In period two, subjects will receive GSK1349572 30mg q24h in combination with ATV 400mg q24h (treatment C) for 14 days. There will be no washout between treatment periods. Day 1 of Period 2 will be the day after Day 5 of Period 1. Subjects will have a screening visit within 30 days prior to the first dose of study drug, two treatment periods, and a follow-up visit 7-14 days after the last dose of study drug.
  Interventions: Drug: GSK1349572; Drug: Atazanavir 400 mg
- Sequence 1 (Experimental): In the first treatment period, all subjects will receive GSK1349572 30mg q24h for 5 days (treatment A). In period two, subjects will receive GSK1349572 30mg q24h in combination with ATV/RTV 300/100mg q24h (treatment B) for 14 days. There will be no washout between treatment periods. Day 1 of Period 2 will be the day after Day 5 of Period 1. Subjects will have a screening visit within 30 days prior to the first dose of study drug, two treatment periods, and a follow-up visit 7-14 days after the last dose of study drug.
  Interventions: Drug: GSK1349572; Drug: Atazanavir 300 mg; Drug: Ritonavir

INTERVENTIONS:
Drug: GSK1349572 — GSK1349572 30 mg once a day for 5 days in Period 1 and 14 days in Period 2
Drug: Atazanavir 300 mg — Atazanavir 300 mg once per day for 14 days in Period 2
  Other Names: ATV; REYATAZ. REYATAZ is a registered trademark of Bristol-Myers Squibb Company
  Arms: Sequence 1
Drug: Atazanavir 400 mg — Atazanavir 400 mg once a day for 14 days in Period 2
  Other Names: REYATAZ. REYATAZ is a registered trademark of Bristol-Myers Squibb Company; ATV
  Arms: Sequence 2
Drug: Ritonavir — Ritonavir 100 mg once a day for 14 days in Period 2
  Other Names: NORVIR. NORVIR is a registered trademark of Abbott Labs; RTV
  Arms: Sequence 1

SUMMARY:
The purpose of this study is to compare the amount of GSK1349572 (study drug) in the blood when given with and without atazanavir/ritonavir or atazanavir and to compare the blood levels of atazanavir when given with GSK1349572 to historical data for atazanavir.

DETAILED DESCRIPTION:
GSK1349572 is an integrase inhibitor that will be evaluated for the treatment of HIV infection. As GSK1349572 progresses into clinical trials in HIV-infected patients where combination antiretroviral therapy is the standard of care, it is likely that it will be dosed with protease inhibitors (PIs) including atazanavir/ritonavir (ATV/RTV) and atazanavir alone. Ritonavir is a substrate of CYP3A and inhibitor of CYP3A and Pgp and atazanavir is an inhibitor of UGT1A1. Ritonavir is also a known inducer of CYP and UGT enzymes. As GSK1349572 likely undergoes metabolism by CYP and UGT enzymes and is a Pgp substrate, a drug interaction study between GSK1349572 and ATV is warranted. GSK1349572 is not an inhibitor or inducer of CYP3A and is not expected to have impact on pharmacokinetics (PK) of atazanavir and ritonavir. Accordingly, the primary objective of this study is to compare steady-state plasma PK, safety and tolerability of GSK1349572 30 mg every 24h (q24h) with and without ATV/RTV 300/100 mg q24h or ATV 400mg q24h.

Approximately 24 subjects will receive GSK1349572 30mg q24h for 5 days (Treatment A). Subjects will then be administered GSK1349572 30mg q24h in combination with either ATV/RTV 300/100 mg q24h (Treatment B, n=12) or ATV 400 mg q24h (Treatment C, n=12) for 14 days. There will be no washout between treatments. Safety evaluations and serial PK samples will be collected during each treatment period. A follow-up visit will occur 7-14 days after the last dose of study drug.

This study will be conducted at one center in the US, with healthy adult male and female subjects.

ELIGIBILITY:
Inclusion Criteria:

* AST, ALT, and alkaline phosphatase less than or equal to 1.5xULN. Total bilirubin must be less than ULN.
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and ECG.
* Male or female between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of: Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation, hysterectomy or bilateral oophorectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/ml and estradiol < 40 pg/ml (<140 pmol/L) is confirmatory].
* Male subjects must agree to use one of the contraception methods listed in the protocol. This criterion must be followed from the time of the first dose of study medication until 14 days post-last dose.
* Body weight greater than or equal to 50 kg for men and greater than or equal to 45 kg for women and body mass index (BMI) within the range 18.0-32.0 kg/m2 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

* The subject has a positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* History of sensitivity to any of the study medications, or components thereof, including sulfa-containing drugs, or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* If heparin is used during PK sampling, subjects with a history of sensitivity to heparin or heparin-induced thrombocytopenia should not be enrolled.
* History of regular alcohol consumption within 6 months of the study defined as: An average weekly intake of >14 drinks/week for men or >7 drinks/week for women. One drink is equivalent to (12 g alcohol) = 5 ounces (150 ml) of wine or 12 ounces (360 ml) of beer or 1.5 ounces (45 ml) of 80 proof distilled spirits.
* Has a history or regular use of tobacco- or nicotine-containing products within 3 months prior to screening.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice from 7 days prior to the first dose of study medication.
* Pregnant females as determined by positive serum or urine human chorionic gonadotrophin (hCG) test at screening or prior to dosing.
* Lactating females.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subjects with a pre-existing condition interfering with normal gastrointestinal anatomy or motility, hepatic and/or renal function, that could interfere with the absorption, metabolism, and/or excretion of the study drugs. Subjects with a history of cholecystectomy, peptic ulceration, inflammatory bowel disease or pancreatitis should be excluded.
* History/evidence of symptomatic arrhythmia, angina/ischemia, coronary artery bypass grafting (CABG) surgery or percutaneous transluminal coronary angioplasty (PCTA) or any clinically significant cardiac disease.
* History/evidence of clinically significant pulmonary disease.
* History of significant renal or hepatobiliary diseases. Subjects with a history of nephrolithiasis will be excluded.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* A positive test for HIV antibody.
* History of 2nd degree or higher AV block.
* History of Gilbert's disease.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* The subject's systolic blood pressure is outside the range of 90-140mmHg, or diastolic blood pressure is outside the range of 45-90mmHg or heart rate is outside the range of 50-100bpm for female subjects or 45-100 bpm for male subjects.
* Dcreening ECG within protocol limits (a single repeat is allowed for eligibility determination)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-04; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Plasma GSK1349572 steady-state AUC(0-tau), Cmax, C0, Ctau, and Cmin following administration of GSK1349572 30mg q24h for 5 days and following co-administration with ATV/RTV 300/100mg q24h or ATV 400mg q24h for 14 days. | 19 days

SECONDARY OUTCOMES:
Safety and tolerability parameters, including adverse event, concurrent medication, clinical laboratory, ECG, and vital signs assessments. | 19 days
Plasma GSK1349572 PK parameters: tmax, tmin, CL/F and t½, following administration of GSK1349572 30mg q24h for 5 days and following co-administration with ATZ/RTV 300/100mg q24h or ATZ 400mg q24h for 14 days. | 19 days
Plasma ATV PK parameters, including AUC(0-tau), Cmax, Ctau, and Cmin following co-administration of GSK1349572 30mg q24h and ATV/RTV 300/100mg q24h or ATV 400mg q24h for 14 days. | 19 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Austin, Texas, United States